CLINICAL TRIAL: NCT00510250
Title: A Phase I/II Study of Cisplatin and Radiation in Combination With Sorafenib in Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDPDRO-002; Bayer Protocol# 12138
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Cancer of the Cervix
Keywords: Cervix Cancer; Cervical Cancer; Sorafenib; Cisplatin; Radiation; Radiotherapy; Phase I; Phase II; Carcinoma; Cancer; Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma; Neoplasms | interventions — Sorafenib; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin and Radiation in Combination with Sorafenib (Experimental)
  Interventions: Drug: Sorafenib; Drug: Cisplatin; Procedure: Radiation

INTERVENTIONS:
Drug: Sorafenib — 200mg PO BID x 7 days prior to Radiation and Cisplatin for Low-Risk Patients or 200mg PO BID x 7 days prior to, and 35 days during Radiation and Cisplatin for High-Risk Patients
Drug: Cisplatin — 40mg/m2 administered weekly via IV, with Radiation
Procedure: Radiation — Administered for 30-40 days.Combination of external beam radiotherapy followed by intra-cavitary brachytherapy.

SUMMARY:
This will be a multi-institution, single-arm, open-label, phase I/II trial. Eligible patients will have pathologically-proven T1b-3b, N0/1, M0 epithelial carcinoma of the cervix. We hypothesize that sorafenib in combination with chemotherapy and radiotherapy may have anti-tumor activity in patients with cervical cancer. Sorafenib has not previously been combined with conventional RT-CT to treat cervix cancer.

DETAILED DESCRIPTION:
During the phase I component of the study, low risk patients (tumor size ≤5 cm and radiographically node negative) will receive sorafenib alone in escalating doses for at least 1 week prior to the start of conventional treatment with radiotherapy and chemotherapy (RT-CT). High risk patients (tumor > 5 cm or node positive) will receive sorafenib alone in escalating dose for at least 1 week prior to the start of RT-CT, as well as concurrently with RT-CT. Cohorts of 3 patients per dose level are planned. If 1/3 patients encounters a dose-limiting toxicity (DLT), then that cohort will be expanded to 6 patients. If >2/3 of patients encounter a DLT, then that dose level will be declared as the maximum tolerated dose (MTD). An additional 3 patients will be entered into the dose level one below the MTD. The recommended phase II dose (RPTD) is defined as the dose level with < 1/6 patients with DLT.

For the phase II component, all patients will receive sorafenib at the RPTD for at least 1 week prior to, and concurrent with, RT-CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-proven epithelial carcinoma of the cervix, T1B-3B, N0/1, M0 with visible or palpable disease and a decision to treat radically with radiotherapy and concurrent cisplatin chemotherapy (RT-CT).
* ECOG performance status 0, 1 or 2 (Karnofsky>=60%)
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes >3,000/mcL
  * Absolute neutrophil count >1,500/mcL
  * Platelets >100,000/mcL
  * Hemoglobin > 9 g/dL
  * Total bilirubin Within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <=2.5 X institutional upper limit of normal
  * Creatinine Within normal institutional limits, or
  * Creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above normal
* No prior treatment for cervix cancer.
* The effects of sorafenib on the developing human fetus at the recommended therapeutic dose are unknown. Although radical RT-CT for cervix cancer is not compatible with survival of a developing fetus, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* No active malignancy at another site.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents concurrently or within 4 weeks. Patients who have previous exposure to a raf-kinase inhibitor are excluded
* Patients with poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher, or diastolic blood pressure of 90 mmHg or higher) are ineligible.
* Patients with any condition that impairs their ability to swallow sorafenib tablets are excluded (e.g. gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease).
* Bleeding disorders. Patients cannot be receiving therapeutic anticoagulation. Prophylactic anticoagulation (ie. low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for PT, INR, or PTT are met.
* Patients with known brain metastases should be excluded because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. These patients would not be eligible for radical RT-CT for cervix cancer, but instead would be treated for palliation.
* Patients with intercurrent cardiac dysfunction including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia are excluded as are those with a history of ischemic heart disease including myocardial infarction.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because sorafenib has the potential for teratogenic or abortifacient effects as shown by the gross fetal malformations and effects on embryo-fetal survival seen in reproductive toxicity studies in the rat. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sorafenib, breastfeeding should be discontinued if the mother is treated with sorafenib.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with sorafenib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* A decision to treat with extended-field pelvic and para-aortic radiotherapy, specifically cases where the para-aortic field will extend cranial to the L3-4 vertebral inter-space.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-06; Primary Completion 2010-09 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Determine the biologic activity of sorafenib in cervix cancer. | Not Determined

SECONDARY OUTCOMES:
Determine the acute and late toxicity, and effect of sorafenib in combination with radiation and chemotherapy on the disease-free survival of patients with high-risk cervix cancer. | Not Determined

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, MD FRCP, Principal Investigator — Princess Margaret Hospital, Canada; Michael Milosevic, MD FRCPC, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada